CLINICAL TRIAL: NCT04942899
Title: Aromatase Inhibitors Plus Metronomic Capecitabine in Treatment of Patients With Recurrent or Metastatic Hormone Receptor Positive, HER2 Negative Breast Cancer
Brief Title: Letrozole Plus Metronomic Capecitabine as First-line Treatment for Patients With Recurrent or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yosra farghaly sayed mahmoud, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AIs with chemotherapy in MBC
Record Dates: First submitted 2021-06-06; First posted 2021-06-29 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Metastasis Breast
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: letrozole — concurrent capecitabine 500 mg three times daily in combination with letrozole 2.5 mg orally once daily.
  Other Names: capecitabine

SUMMARY:
The study is designed to assess the treatment outcomes following treatment with letrozole plus metronomic capecitabine in patients with hormone receptor-positive, Her2-negative advanced breast cancer who have not received prior systemic anti-cancer therapies for their recurrent /metastatic disease.

DETAILED DESCRIPTION:
Breast cancer is recognized as the commonest cancer in females, and the second commonest malignant tumor, after lung cancer, in overall figures worldwide.

In 2021, an estimated 281,550 new cases of invasive breast cancer are expected to be diagnosed in women in the U.S., along with 49,290 new cases of non-invasive (in situ) breast cancer.

About 43,600 women in the U.S. are expected to die in 2021 from breast cancer. Death rates have been steady in women under 50 since 2007, but have continued to drop in women over 50. The overall death rate from breast cancer decreased by 1% per year from 2013 to 2018. These decreases are thought to be the result of treatment advances and earlier detection through screening.

According to the World Health Organization, breast cancer became the most common cancer globally as of 2021, accounting for 12% of all new annual cancer cases worldwide.

Breast cancer is increasingly recognized as a heterogeneous disease exhibiting substantial differences concerning biological behavior and requiring distinct therapeutic interventions. There has been a continuous decline in mortality over recent years due to improvements in early diagnosis and the increased availability of more effective treatments. However, despite these improvements, The treatment of hormone receptor-positive metastatic breast cancer (MBC) who developed disease progression on first-line hormonal treatment that included aromatase inhibitors (AI) represents a challenge as those patients ultimately develop resistant disease unresponsive to standard lines of estrogen receptors (ER) blockade. Capecitabine is an oral chemotherapy that mimics continuous infusion of 5-FU with known activity in MBC. It might be preferred because of its tolerability and relatively lower toxicity than other chemotherapeutic agents. Metronomic chemotherapy is defined as the frequent (daily, many times a week, or weekly) or continuous administration of low dose chemotherapeutic agents, without prolonged drug-free intervals. This way of administration improves the antiangiogenic activity of chemotherapy. Another important advantage of this approach is the significant reduction in toxicity. Capecitabine's pharmacokinetics and high safety profile make it a suitable drug for metronomic administration. Many studies reported that the overall response rate can be improved by (15.8-21.7%) when metronomic chemotherapy is combined with aromatase inhibitors. This combination can also decrease the level of both the Ki-67 index and VEGF-A significantly in the tumor tissue. It was reported that the patients who received letrozole plus metronomic chemotherapy achieved a higher overall response rate (ORR) than those who received letrozole alone (87.7% vs 71.9% respectively.

ELIGIBILITY:
Inclusion Criteria:

* Female patients > 18 years old with loco regionally recurrent or metastatic disease not amenable to curative therapy
* Confirmed diagnosis of hormonal receptor positive (HR+)/Her2-negative breast cancer
* If the patient is pre-/peri- menopausal, a luteinizing hormone releasing hormone (LHRH) agonist will be given for at least 28 days before randomization or ovarian ablation or suppression by surgery or radiotherapy
* Measurable disease defined by RECIST version 1.1,
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Adequate organ and marrow function

Exclusion Criteria:

* Patients with advanced, symptomatic visceral spread (visceral crisis)
* Patients diagnosed with central nervous system metastases
* Second primary malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
tumor response | 1 year
  tumor response in form of change tumor size

SECONDARY OUTCOMES:
progression free survival | 1 year
  decrease sites of metastasis

REFERENCES:
- [Background] Shankar A, Rath G, Roy S, Malik A, Bhandari R, Kishor K, Barnwal K, Upadyaya S, Srivastava V, Singh R. Level of awareness of cervical and breast cancer risk factors and safe practices among college teachers of different states in india: do awareness programmes have an impact on adoption of safe practices? Asian Pac J Cancer Prev. 2015;16(3):927-32. doi: 10.7314/apjcp.2015.16.3.927. PMID 25735384
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of chemotherapy and hormonal therapy for early breast cancer on recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 May 14-20;365(9472):1687-717. doi: 10.1016/S0140-6736(05)66544-0. PMID 15894097
- [Background] Winkfield KM, Harris JR. Effective local therapy and long-term survival in breast cancer. Oncology (Williston Park). 2009 Jul;23(8):669-75. PMID 19711579
- [Background] Schwartzberg LS, Wang G, Somer BG, Blakely LJ, Wheeler BM, Walker MS, Stepanski EJ, Houts AC. Phase II trial of fulvestrant with metronomic capecitabine for postmenopausal women with hormone receptor-positive, HER2-negative metastatic breast cancer. Clin Breast Cancer. 2014 Feb;14(1):13-9. doi: 10.1016/j.clbc.2013.09.003. Epub 2013 Sep 27. PMID 24268206
- [Background] Van Cutsem E, Twelves C, Cassidy J, Allman D, Bajetta E, Boyer M, Bugat R, Findlay M, Frings S, Jahn M, McKendrick J, Osterwalder B, Perez-Manga G, Rosso R, Rougier P, Schmiegel WH, Seitz JF, Thompson P, Vieitez JM, Weitzel C, Harper P; Xeloda Colorectal Cancer Study Group. Oral capecitabine compared with intravenous fluorouracil plus leucovorin in patients with metastatic colorectal cancer: results of a large phase III study. J Clin Oncol. 2001 Nov 1;19(21):4097-106. doi: 10.1200/JCO.2001.19.21.4097. PMID 11689577
- [Background] Seidman AD, O'Shaughnessy J, Misset JL. Single-agent capecitabine: a reference treatment for taxane-pretreated metastatic breast cancer? Oncologist. 2002;7 Suppl 6:20-8. doi: 10.1634/theoncologist.7-suppl_6-20. PMID 12454316
- [Background] Walko CM, Lindley C. Capecitabine: a review. Clin Ther. 2005 Jan;27(1):23-44. doi: 10.1016/j.clinthera.2005.01.005. PMID 15763604
- [Background] Munzone E, Di Pietro A, Goldhirsch A, Minchella I, Verri E, Cossu Rocca M, Marenghi C, Curigliano G, Radice D, Adamoli L, Nole F. Metronomic administration of pegylated liposomal-doxorubicin in extensively pre-treated metastatic breast cancer patients: a mono-institutional case-series report. Breast. 2010 Feb;19(1):33-7. doi: 10.1016/j.breast.2009.10.003. Epub 2009 Nov 1. PMID 19884008
- [Background] Mehta RS. Dose-dense and/or metronomic schedules of specific chemotherapies consolidate the chemosensitivity of triple-negative breast cancer: a step toward reversing triple-negative paradox. J Clin Oncol. 2008 Jul 1;26(19):3286-8; author reply 3288. doi: 10.1200/JCO.2008.17.1116. No abstract available. PMID 18591566
- [Background] Emmenegger U, Kerbel RS. Five years of clinical experience with metronomic chemotherapy: achievements and perspectives. Onkologie. 2007 Dec;30(12):606-8. doi: 10.1159/000111479. Epub 2007 Nov 30. No abstract available. PMID 18063872
- [Background] Bottini A, Generali D, Brizzi MP, Fox SB, Bersiga A, Bonardi S, Allevi G, Aguggini S, Bodini G, Milani M, Dionisio R, Bernardi C, Montruccoli A, Bruzzi P, Harris AL, Dogliotti L, Berruti A. Randomized phase II trial of letrozole and letrozole plus low-dose metronomic oral cyclophosphamide as primary systemic treatment in elderly breast cancer patients. J Clin Oncol. 2006 Aug 1;24(22):3623-8. doi: 10.1200/JCO.2005.04.5773. PMID 16877730
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437